CLINICAL TRIAL: NCT01696708
Title: Study of the Brain Energy Profile Evolution, Using 31Phosphorus-Nuclear Magnetic Resonance Spectroscopy, at Different Stages of Huntington Disease
Brief Title: Utilization of 31P-Nuclear Magnetic Resonance Spectroscopy to Monitor Brain Energy Deficit in Huntington Disease
Acronym: PRO-MH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C12-49; 2012-A01063-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-20; First posted 2012-10-01 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2012-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): 31-Phosphorus RMN Spectroscopy
  Interventions: Other: 31-Phosphorus RMN Spectroscopy
- Volunteers (Other): 31-Phosphorus RMN Spectroscopy
  Interventions: Other: 31-Phosphorus RMN Spectroscopy

INTERVENTIONS:
Other: 31-Phosphorus RMN Spectroscopy

SUMMARY:
The purpose of this project is to study brain energy profile evolution at different stages of the Huntington disease.

ELIGIBILITY:
Inclusion Criteria:

* UHDRS < 50
* Age > 18 years
* Ability to undergo MR scanning
* Covered by french social security

Exclusion Criteria:

* Evidence of psychiatric disorder
* Attendant neurological disorder
* Contraindications to MRI (claustrophobia, metallic or material implants)
* Severe head injury
* Unable to understand the protocol
* Pregnancy
* Failure to give informed consent
* Subjects with exclusion criteria required by french law (e.g. subjects who require a legally authorized representative to obtain consent)
* Unwillingness to be informed in case of abnormal MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Ratio of Inorganic Phosphate (Pi) over phosphocreatine (PCr): Pi/PCr | 2 years
  31P-MRS allows quantification of high-energy phosphate metabolites such as phosphocreatine and inorganic phosphate

SECONDARY OUTCOMES:
Correlation between primary outcome measure and clinical parameters | 2 years
  Correlating a brain energy deficit with clinical parameters in Huntington patients such as the Unified Huntington's disease rating scale (UHDRS) and total functional capacity score (TFC).
Study of longitudinal changes in Pi/PCr ratio over time. | 2 years
  Patients will be retested after one month.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Mochel, MD, PhD, Principal Investigator — INSERM UMR S975 Institut du Cerveau et de la Moelle, AP-HP Département de Génétique, Université Pierre et Marie Curie, Paris France
Locations (1):
- Brain and Spine Institute (ICM), Paris, France

REFERENCES:
- [Result] Adanyeguh IM, Monin ML, Rinaldi D, Freeman L, Durr A, Lehericy S, Henry PG, Mochel F. Expanded neurochemical profile in the early stage of Huntington disease using proton magnetic resonance spectroscopy. NMR Biomed. 2018 Mar;31(3):10.1002/nbm.3880. doi: 10.1002/nbm.3880. Epub 2018 Jan 9. PMID 29315899
- [Result] Adanyeguh IM, Rinaldi D, Henry PG, Caillet S, Valabregue R, Durr A, Mochel F. Triheptanoin improves brain energy metabolism in patients with Huntington disease. Neurology. 2015 Feb 3;84(5):490-5. doi: 10.1212/WNL.0000000000001214. Epub 2015 Jan 7. PMID 25568297